CLINICAL TRIAL: NCT02883465
Title: Ultrasound Diagnostic for Diaphragmatic Dysfunction in Reanimation and Influence Over Mechanical Ventilation Weaning Period
Brief Title: Ultrasound Diagnostic for Diaphragmatic Dysfunction in Reanimation
Acronym: ECHODIAPH II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other)
Collaborators: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SJSL12014
Record Dates: First submitted 2016-05-27; First posted 2016-08-30 (Estimated); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Mechanical Ventilation Weaning
Keywords: diaphragmatic dysfunction; mechanical ventilation weaning; failure extubation rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Other)
  Interventions: Procedure: Diaphragmatic ultrasound

INTERVENTIONS:
Procedure: Diaphragmatic ultrasound — All patients will have a diaphragmatic ultrasound in the 4 hours before the extubation.
  * a record of the right and left diaphragmatic cupolas run, with a chest approach and using a 4-5 MHz (megahertz) cardiac or abdominal sensor. 3 acquisitions for each side
  * a record of the diaphragm thickening at the right and left apposition zones with a 10-12 MHz (megahertz) vascular sensor. 3 acquisitions for each side

SUMMARY:
Extubation is a crucial step when patients are being weaned from mechanical ventilator support. Indeed, the patient has to face an increasing burden imposed to the ventilation system. The ability to overcome this event will determine the patient survival. A warning signal could be very useful is this situation. 2 recent studies have shown that measuring diaphragmatic cupolas and muscular fibers thickening fraction could help to spot a population with a high risk of "diaphragmatic weakness", characterized by a high failure extubation rate. This study aims to verify that this kind of group of patients does exist.

ELIGIBILITY:
Inclusion Criteria:

* Successful spontaneous breathing trial and extubation expected on the same day and 1 of the following criteria :
* Age > 65
* Mechanical ventilation during > 7 days
* Cardiac history (ischemic, rhythmic or valve cardiopathy)
* Respiratory history (documented or likely chronic respiratory failure)

Exclusion Criteria:

* Patient who is tracheotomized
* Peripheric neuromuscular disease (myasthenia, myopathy)
* Surgery circumstances that could affect the quality of the ultrasound exam (drains or bandages)
* Pregnant woman
* Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-03-06 (Actual); Primary Completion 2016-10-28 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Extubation success rate | 7 days after the reported extubation
  Extubation success rate, defined as no reintubation 7 days after the reporting extubation

SECONDARY OUTCOMES:
Length of stay in reanimation unit (days) | At discharge of reanimation unit (up to 1 year)
Length of mechanical ventilation | At the extubation time
Number of patients with invasive or non-invasive mechanical ventilation | 48 hours after the extubation
  Resort to invasive or non-invasive mechanical ventilation
Mortality | At discharge of reanimation unit (up to 1 year)
Comparison between the predictive value of diaphragmatic ultrasound dysfunction and a clinical parameter : cough strength measured with a defined scale | At the extubation time
  The scale used to measure the cough is the following :
  * absent
  * inefficient
  * low efficiency
  * mild efficiency
  * efficient
Comparison between the predictive value of diaphragmatic ultrasound dysfunction and a clinical parameter : quantity of secretions measured with a defined scale | At the extubation time
  * any secretions
  * low secretions
  * mild secretions
  * abundant secretions
  * very abundant secretions
Comparison between the predictive value of diaphragmatic ultrasound dysfunction and a clinical parameter : presence/absence or cervical tonus | At the extubation time
Comparison between the predictive value of diaphragmatic ultrasound dysfunction and a clinical parameter : F/Vt ratio measured in breaths/min/L | At the extubation time
Comparison between the predictive value of diaphragmatic ultrasound dysfunction and a paraclinical parameter : maximal inspiratory pressure in centimeters of water | At the extubation time
Comparison between the predictive value of diaphragmatic ultrasound dysfunction and a paraclinical parameter : minimal expiratory pressure measured in centimeters of water | At the extubation time
Comparison between the predictive value of diaphragmatic ultrasound dysfunction and a paraclinical parameter : peak flow measured in L/min (liters per minute) | At the extubation time
Comparison between the predictive value of diaphragmatic ultrasound dysfunction and a paraclinical parameter : peak flow when coughing measured in L/min (liters per minute) | At the extubation time
Comparison between the predictive value of diaphragmatic ultrasound dysfunction and a paraclinical parameter : P0,1 measured in milliseconds | At the extubation time

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre Hospitalier Saint Joseph Saint Luc, Lyon
  - Centre Hospitalier Annecy Genevois, Metz-Tessy
  - Centre Hospitalier Universitaire de Poitiers, Poitiers